CLINICAL TRIAL: NCT01634230
Title: Emergency Use of OCR-002 (Ornithine Phenylacetate) in the Treatment of Patients With Acute Liver Failure
Brief Title: Emergency Use of OCR-002 in Acute Liver Failure (ALF)
Status: No longer available | Type: Expanded Access
Sponsor: Ocera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Other Study IDs: OCR002-EmUse-001
Record Dates: First submitted 2012-06-25; First posted 2012-07-06 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — ornithine phenylacetate

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: OCR-002 — daily dose: 10 g infused over 24 hours
  Other Names: ornithine phenylacetate

SUMMARY:
This study provides emergency use of the unapproved study medication in ALF patients with acute liver failure who are not responding to standard of care.

DETAILED DESCRIPTION:
This is an open-label study in patients diagnosed with ALF who are not responding to the institution's standards of care. Standard of care may include, but is not limited to, administration of N-acetylcysteine, lactulose, hypothermia therapy, and consideration for orthotopic liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* International Normalized Ratio (INR) ≥1.5 with encephalopathy in patient with no prior history of liver disease
* Venous ammonia level of ≥ 100 μmol/L

Exclusion Criteria:

* Patients who are pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Ocera Therapeutics
Locations (1):
- University of Arkansas, Little Rock, Arkansas, United States